CLINICAL TRIAL: NCT03468244
Title: Clinical Study of Personalized mRNA Tumor Vaccine Encoding Neoantigen in Patients With Advanced Esophageal Squamous Carcinoma, Gastric Adenocarcinoma, Pancreatic Adenocarcinoma and Colorectal Adenocarcinoma
Brief Title: Clinical Study of Personalized mRNA Vaccine Encoding Neoantigen in Patients With Advanced Digestive System Neoplasms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: Stemirna Therapeutics (Industry)
Responsible Party: Principal Investigator, Bin Wang, Attending physician, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHO-01002
Record Dates: First submitted 2018-03-08; First posted 2018-03-16 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Advanced Esophageal Squamous Carcinoma; Gastric Adenocarcinoma; Pancreatic Adenocarcinoma; Colorectal Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized mRNA Tumor Vaccine (Experimental): Personalized mRNA Tumor Vaccine Encoding Neoantigen in Patients with Advanced Esophageal Squamous Carcinoma, Gastric Adenocarcinoma, Pancreatic Adenocarcinoma and Colorectal Adenocarcinoma
  Interventions: Biological: Personalized mRNA Tumor Vaccine

INTERVENTIONS:
Biological: Personalized mRNA Tumor Vaccine — subcutaneous injection with personalized mRNA tumor vaccine at least four times

SUMMARY:
A single arm, open-label pilot study is designed to determine the safety, tolerability and effectiveness of personalized mRNA tumor vaccine encoding neoantigen in Patients with advanced esophageal squamous carcinoma, gastric adenocarcinoma, pancreatic adenocarcinoma and colorectal adenocarcinoma

DETAILED DESCRIPTION:
Dr. Bin Wang developed the investigational vaccine used in this clinical trial and designed the trial protocol.For patients with advanced esophageal squamous carcinoma, gastric adenocarcinoma, pancreatic adenocarcinoma and colorectal adenocarcinoma tumor who have disease progression with first line chemotherapy. Single or multiple doses of personalized mRNA tumor vaccine encoding neoantigen will be given to observe the safety and efficacy the mRNA tumor vaccine.

Primary objectives:

Determine the safety, tolerability and cytokinetics of the personalized mRNA tumor vaccine in patients with advanced esophageal squamous carcinoma, gastric adenocarcinoma, pancreatic adenocarcinoma and colorectal adenocarcinoma.

Secondary objectives:

Make a preliminary evaluation on the efficacy of personalized mRNA tumor vaccine in patients with advanced esophageal squamous carcinoma, gastric adenocarcinoma, pancreatic adenocarcinoma and colorectal adenocarcinoma with the following parameters:

Time of tumor progression (TTP);

Disease Control Rate (DCR);

Objective Remission Rate (ORR);

Overall Survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 - 75 with pathologically confirmed advanced Esophageal Squamous Carcinoma, Gastric Adenocarcinoma, Pancreatic Adenocarcinoma and Colorectal Adenocarcinoma.
2. Patients with advanced Esophageal Squamous Carcinoma, Gastric Adenocarcinoma, Pancreatic Adenocarcinoma and Colorectal Adenocarcinoma who have disease progression with first line chemotherapy. (1) Failure of treatment is defined as disease progression, recurrence or metastatic disease, or intolerable toxicities occurred after treatment. (2) Each line of treatment during the period of disease progression includes one or more chemotherapy drugs which are administered for not less than one cycle or even longer. Neoadjuvant/adjuvant therapy can be applied at an earlier stage of treatment. If patient has developed recurrence or metastatic disease within 24 weeks of neoadjuvant/adjuvant therapy, it is considered as one line of systemic chemotherapy. (3) Therapies that can be performed at an earlier stage are chemotherapy in conjunction with molecular targeted drugs.
3. Expected survival after first dose of study drug > 24 weeks.
4. At least one measurable lesion (≥ 10 mm) for imaging assessment.
5. ECOG scores 0 - 1.
6. Fresh pathological tissue specimens can be obtained
7. White blood cells (WBCs) ≥ 2.5×10^9/L

   * Platelets (PLT) ≥ 100×10^9/L
   * Hemoglobin, Blood (Hb) ≥ 9.0 g/dL
   * MID ≥ 1.5×10^9/L
   * Lymphocyte (LY) ≥ 0.47×10^9/L
   * LY% ≥ 15%
8. Serum albumin (Alb) ≥ 30 g/L
9. Serum lipase (LPS) and serum amylase < 1.5 ULN
10. Serum creatinine ≤ 1.5 ULN
11. Alanine aminotransferase (ALT) ≤ 2.5 ULN

    * Aspartate aminotransferase (AST) ≤ 2.5 ULN
    * If osseous metastasis or liver metastasis is developed and alkaline phosphatase • (ALP) > 2.5 ULN, ALT and AST < 1.5 ULN.
12. Serum total bilirubin (TBIL) ≤ 1.5 ULN
13. Prothrombin Time (PT): International Normalized Ratio (INR) < 1.7.

    * PT < (ULN + 4) s

All test results should be within their normal ranges, and the patient is not receiving continuous supportive care.

Exclusion Criteria:

Patients with any of the following conditions are not eligible for the study.

1. Pregnant or lactating women.
2. HIV positive, HCV positive, HBV DNA copies ≥ 10^3.
3. Uncontrolled active infection.
4. Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary.
5. Allergic to immunotherapies and related drugs.
6. Untreated brain metastases or having symptoms of brain metastases.
7. Metastases to the lung: central tumor or multiple metastases.
8. Patients with heart disease for which treatment is needed or with poorly controlled hypertension.
9. Patients with unstable or active peptic ulcer or with alimentary tract hemorrhage.
10. Patients with previous organ transplantation or in preparation for organ transplantation.
11. Patients have undertaken major surgeries or have been badly injured 4 weeks before the study (blood collection), or will undertake major surgeries during the study.
12. The judgment of investigators that the patient is not able to or not willing to follow the instructions of the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 24 weeks
  During the trial conduction, especially within the 24 weeks of treatment phase when mRNA tumor Vaccine administered, all adverse events (including laboratory abnormality and clinical events) will be closely monitored, and all ≥ grade 3 adverse events per CTCAE (v 3.0) will be recorded, including but not limited to the toxicities potentially suspected to relate to injection procedures and/or mRNA Tumor Vaccine therapy as listed below:
  * Fever
  * Chills
  * Nausea, vomiting and other gastrointestinal symptoms
  * Fatigue
  * Hypotension
  * Respiratory distress
  * Tumor lysis syndrome
  * Neutropenia, thrombocytopenia
  * Liver and kidney dysfunction

SECONDARY OUTCOMES:
Disease Control Rate of Personalized mRNA Tumor Vaccine | 1.5 years
  Disease Control Rate (DCR)
Progression-free Survival of Personalized mRNA Tumor Vaccine | 2 years
  Progression-free Survival (PFS)
Time to Tumor Progression of Personalized mRNA Tumor Vaccine | 2 years
  Time to Tumor Progression (TTP)
Overall Survival of Personalized mRNA Tumor Vaccine | 3 years
  Overall Survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Xianbao Zhan, Dr., Study Director — Chanhai hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang B, Peng X, Li J, Wang Y, Chen L, Wu M, Zhang Y, Wang W, Feng D, Tang S, Zhang L, Zhan X. Personalized mRNA vaccine combined with PD-1 inhibitor therapy in a patient with advanced esophageal squamous cell carcinoma. Am J Cancer Res. 2024 Aug 25;14(8):3896-3904. doi: 10.62347/NVFB3780. eCollection 2024. PMID 39267685